CLINICAL TRIAL: NCT00003476
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Children With Primary Malignant Brain Tumors
Brief Title: Antineoplaston Therapy in Treating Children With Primary Malignant Brain Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066513; BC-BT-22 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Childhood Brain Tumor
Keywords: childhood anaplastic astrocytoma; recurrent childhood anaplastic astrocytoma; childhood glioblastoma multiforme; recurrent childhood glioblastoma multiforme; childhood brainstem glioma; recurrent childhood brainstem glioma; childhood primitive neuroectodermal tumor; recurrent childhood primitive neuroectodermal tumor
MeSH Terms: conditions — Astrocytoma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Children with a primary malignant brain tumor will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for children with primary malignant brain tumors provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of children with primary malignant brain tumors.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on children with primary malignant brain tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in children with primary malignant brain tumors as measured by an objective response to therapy (complete response, partial response) or stable disease.
* To determine the safety and tolerance of Antineoplaston therapy in children with primary malignant brain tumors.

OVERVIEW: This is a single arm, open-label study in which children with primary malignant brain tumors receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed incurable primary malignant brain tumor that has progressed, recurred, or persisted after initial therapy (must have failed standard therapy).
* Evidence of residual tumor by MRI performed within two weeks prior to study entry

PATIENT CHARACTERISTICS:

Age:

* 6 months to 17 years

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* WBC at least 1,500/mm^3
* Platelet count greater than 50,000/mm^3

Hepatic:

* No hepatic failure
* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal

Renal:

* Creatinine no greater than 2.5 mg/dL

Cardiovascular:

* No severe heart disease
* No uncontrolled hypertension

Pulmonary:

* No severe lung disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study participation
* No serious active infections or fever
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulating agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Recovered from prior endocrine therapy
* Concurrent corticosteroids for cerebral edema allowed

Radiotherapy:

* At least 8 weeks since prior radiotherapy (unless clear radiological evidence of progression) and recovered

Surgery:

* At least 4 weeks since prior surgery (unless clear radiological evidence of progression) and recovered

Other:

* No prior antineoplaston therapy

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 1996-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burzynski SR, Janicki TJ, Burzynski GS, Marszalek A, Brookman, S. A phase II study of Antineoplastons A10 and AS2-1 in children with recurrent, refractory or progressive primary brain tumors - Final Report (Protocol BT-22). Journal of Cancer Therapy, 5:977-988, 2014.
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight patients were recruited between March 1966 and November 2011. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 8
Completed | 7
Not Completed | 1
Not completed — Not evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: Years] | 9.1 [2.6 to 16.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks; Stable Disease (SD), <50% decrease and <25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least eight weeks; Progressive Disease (PD), >=25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 7
Participants
  Partial Response | 1
  Stable Disease | 1
  Progressive Disease | 5

2. Secondary Outcome: Percentage of Participants Who Survived
Description: Six months and Twelve months overall survival
Time Frame: 6 months, 12 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 8
Percentage of participants
  6 months overall survival | 50.0
  12 months overall survival | 0

ADVERSE EVENTS:
Time Frame: 15 years, 10 months
Description: Eight patients were recruited between March 1996 and November 2011. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 2/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=8)
Central venous catheter: Thrombosis/embolism (General disorders) | 1 — The Central venous catheter: Thrombosis/embolism was not related to Antineoplaston therapy.
Fever (General disorders) | 1 — The Fever was not related to Antineoplaston therapy.
Vomiting (Gastrointestinal disorders) | 1 — The Vomiting was not related to Antineoplaston therapy.
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1 — The Infection (documented clinically): Lung (pneumonia) was not related to Antineoplaston therapy.
Hydrocephalus (Nervous system disorders) | 1 — The Hydrocephalus was not related to Antineoplaston therapy.
Seizure (Nervous system disorders) | 1 — The Seizure was not related to Antineoplaston therapy.
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 — The Aspiration was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=8)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 2
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 3
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Central venous catheter: Thrombosis/embolism (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3
Fever (General disorders) | 4
Rigors/chills (General disorders) | 1
Weight gain (General disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Cushingoid appearance (Endocrine disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 2
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Infection (documented clinically): Conjunctiva (Infections and infestations) | 1
Infection (documented clinically): Lung (pneumonia) (Infections and infestations) | 1
Infection (documented clinically): Mucosa (Infections and infestations) | 1
Infection (documented clinically): Sinus (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Sinus (Infections and infestations) | 1
Alkaline phosphatase (Investigations) | 2
Bicarbonate, serum-low (Investigations) | 1
GGT (gamma-Glutamyl transpeptidase) (Investigations) | 1
Hyperchloremia (Investigations) | 1
Hypercholesteremia (Infections and infestations) | 1
Hyperglycemia (Investigations) | 1
Hypernatremia (Investigations) | 1
Hypocalcemia (Investigations) | 1
Hypoglycemia (Investigations) | 1
Hypokalemia (Investigations) | 8
Hypomagnesemia (Investigations) | 2
Metabolic/Laboratory - Other (Investigations) | 1
Uric acid, serum-high (hyperuricemia) (Investigations) | 1
Apnea (Nervous system disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Neuropathy - motor (Nervous system disorders) | 1
Neuropathy: CN III Pupil, upper eyelid, extra ocular movements (Nervous system disorders) | 1
Neuropathy: cranial: CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 1
Neuropathy: cranial: CN VII Motor-face; Sensory-taste (Nervous system disorders) | 1
Neuropathy: cranial: CN VIII Hearing and balance (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 6
Speech impairment (Nervous system disorders) | 1
Diplopia (Eye disorders) | 1
Vision-blurred vision (Eye disorders) | 1
Pain: Head/headache (Nervous system disorders) | 3
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No